CLINICAL TRIAL: NCT00868309
Title: A Comparison of Anavip and CroFab in the Treatment of Subjects With Crotalinae (Pit Viper) Envenomation: A Randomized, Prospective, Open-Label, Controlled, Comparative, Multicenter Study
Brief Title: A Comparison of Crotalinae Equine Immune F(ab)2 Antivenom (Anavip) and Crotalidae Polyvalent Immune Fab,
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN-03/02; AN-03/02 (Other: Bioclon)
Record Dates: First submitted 2008-11-06; First posted 2009-03-24 (Estimated); Results first posted 2009-03-24 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Snake Bite; Blood Coagulation Disorders
Keywords: Snake Bite; Venom and antivenom kinetics
MeSH Terms: conditions — Snake Bites; Blood Coagulation Disorders | interventions — anavip; Crotalidae Polyvalent immune Fab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anavip (Experimental): The initial dose of study drug was administered in a total volume of 500 mL (initial doses only) IV over 30 minutes for Anavip
  Interventions: Biological: Anavip
- CroFab (Active Comparator): The initial dose of study drug was administered in a total volume of 500 mL (initial doses only) IV over 60 minutes for CroFab, or as permitted by IV access.
  Interventions: Biological: CroFab

INTERVENTIONS:
Biological: Anavip — Anavip, 10 vials Intravenous (IV) every 2 hours until initial control has been achieved; then 3 maintenance doses of 4 vials every 6 hrs
  Other Names: Antivenin Crotalinae (pit viper) equine immune F(ab)2
  Arms: Anavip
Biological: CroFab — CroFab, 5 vials Intravenous (IV) every 2 hours until initial control has been achieved; then 3 maintenance doses of 2 vials every 6 hrs
  Arms: CroFab

SUMMARY:
This phase II study was a prospective, randomized, open-label, multi-center study in the United States, involving patients from 18 to 70 years of age, comparing Anavip (Antivenin Crotalinae [pit viper] equine immune F(ab)2; Instituto Bioclon, Mexico City, Mexico) against CroFab (Protherics Inc., Nashville, Tennessee), the only currently approved product for treatment of Crotalinae (pit viper) envenomation in the US.

The study was designed to evaluate the hypothesis that lasting correction of snakebite induced thrombocytopenia and hypofibrinogenemia are possible following correction with F(ab)2 antivenom, by analyzing in detail the relationships among platelet count, fibrinogen, venom levels, and antivenom levels in subjects presenting with thrombocytopenia following crotaline viper envenomation. In the study we expected to see a fall in platelet count following Fab treatment, commensurate with that reported in the past. We hypothesized that following F(ab)2 treatment there would be a slower drop in post-treatment platelet counts, with a relatively higher platelet count at any given point in the follow-up period. We further hypothesized that an initial rise and later fall in platelet count would correspond with rise and fall in antivenom levels, and would be mirrored by concurrent drop and rise in levels of unbound circulating venom.

DETAILED DESCRIPTION:
The overall objective of this Phase 2 open-label comparative study was to demonstrate that the F(ab)2 antivenom Anavip has significantly longer plasma persistence than does Fab, and that this is associated with a slower rise in venom levels and slower decline in platelet count and fibrinogen following hospital discharge of envenomated subjects. The effectiveness of F(ab)2 in preventing the recurrence of coagulopathies after the subject's discharge from hospital will indicate that, inherently, F(ab)2 antivenom has an improved safety profile relative to the Fab antivenom CroFab in treating envenomation by crotaline vipers.

Each subject was assessed for quantitative serum venom levels. Relatively few historical data exist to support the use of venom levels as a surrogate endpoint in envenomation. However, changes in venom levels have been correlated with coagulopathic effects, during both the acute phase of venom toxicity and the post treatment period of recurrent venom effect. Validation of this surrogate endpoint via correlation of venom effect with platelet count and fibrinogen level in this phase II study is intended to support future studies.

The secondary endpoints were the determination of coagulation abnormalities during the follow up period.

ELIGIBILITY:
Inclusion Criteria:

* men and women 18 to 70 years of age
* presenting for emergency treatment of pit viper bite
* informed consent document read and signed by subject

Exclusion Criteria:

* allergy to horse serum, sheep serum, or papaya
* current use of any antivenom, or use within the last month
* current participation in a clinical drug study, or participation within the last month
* pregnancy or breast-feeding
* underlying medical conditions that significantly alter blood coagulation: thrombocytopenia, hemophilia, familial dysfibrinogenemia, leukemia, recent ingestion of superwarfarin compounds (rat poison)
* use of any medication expected to affect platelet count, coagulation factors, or fibrinogen: chemotherapeutic agents, warfarin, heparin, aspirin
* No clinical indications of snake bite envenomation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-01; Primary Completion 2006-08 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter García, MD, Study Director — Instituto Bioclon; Leslie Boyer, MD, Principal Investigator — University of Arizona; Alejandro Alagón, MD, PhD, Principal Investigator — Instituto de Biotecnología UNAM
Locations (1):
- Tucson snakebite investigational site, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects arriving at participating centers with a pit viper bite were evaluated with respect to the inclusion/exclusion criteria.
Groups:
- Anavip Crotalinae (Pit Viper) Equine Immune F(ab)2 Antivenom: Anavip, 10 vials IV every 2 hours until initial control has been achieved; then 3 maintenance doses of 4 vials every 6 hrs
- CroFab Crotalidae Polyvalent Immune Fab, Ovine Antivenom: CroFab, 5 vials IV every 2 hours until initial control has been achieved; then 3 maintenance doses of 2 vials every 6 hrs
Period: Overall Study
Arm/Group | Anavip Crotalinae (Pit Viper) Equine Immune F(ab)2 Antivenom | CroFab Crotalidae Polyvalent Immune Fab, Ovine Antivenom
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anavip Crotalinae (Pit Viper) Equine Immune F(ab)2 Antivenom | CroFab Crotalidae Polyvalent Immune Fab, Ovine Antivenom | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (4.8) | 40.7 (16.5) | 45.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Detection of Plasma Venom Levels During the Post Acute Treatment Period.
Time Frame: Follow up after Maintenance doses were completed. Two Weeks.
Measure: Number; unit: participants
Arm/Group | Anavip Crotalinae (Pit Viper) Equine Immune F(ab)2 Antivenom | CroFab Crotalidae Polyvalent Immune Fab, Ovine Antivenom
Number analyzed (Participants) | 6 | 6
participants
  Detectable venom | 0 | 4
  Undetectable venom | 6 | 2

2. Secondary Outcome: >50,000 Platelets/mm3
Description: Thrombocytopenia during follow up period. Two weeks
Time Frame: Follow up after maintenance dose
Measure: Number; unit: participants
Arm/Group | Anavip Crotalinae (Pit Viper) Equine Immune F(ab)2 Antivenom | CroFab Crotalidae Polyvalent Immune Fab, Ovine Antivenom
Number analyzed (Participants) | 6 | 6
participants
  Thrombocytopenia present | 0 | 3
  Thrombocytopenia absent | 6 | 3

ADVERSE EVENTS:
Arm/Group | Anavip Crotalinae (Pit Viper) Equine Immune F(ab)2 Antivenom | CroFab Crotalidae Polyvalent Immune Fab, Ovine Antivenom
Serious Adverse Events (participants affected / at risk) | 0 | 1
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Anavip Crotalinae (Pit Viper) Equine Immune F(ab)2 Antivenom | CroFab Crotalidae Polyvalent Immune Fab, Ovine Antivenom
Rehospitalization for treatment of thrombocytopenia (Blood and lymphatic system disorders) | 0/6 (0) | 1/6 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anavip Crotalinae (Pit Viper) Equine Immune F(ab)2 Antivenom (N=6) | CroFab Crotalidae Polyvalent Immune Fab, Ovine Antivenom (N=6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Puncture site hemorrhage (General disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
axillary pain (General disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
hypoaesthesia (General disorders) | 1 (1) | 0 (0)
migraine (Nervous system disorders) | 0 (0) | 1 (1)
burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
tremor (Nervous system disorders) | 0 (0) | 1 (1)
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
body temperature increased (Investigations) | 0 (0) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
genital pruritus female (Reproductive system and breast disorders) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less